CLINICAL TRIAL: NCT02488057
Title: Improving Beta Cell Function in Mexican American Women With Prediabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, David Bradley MD, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014H0478
Record Dates: First submitted 2015-06-11; First posted 2015-07-02 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Pre-Diabetes
MeSH Terms: conditions — Glucose Intolerance | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet-induced weight loss (Active Comparator): Investigators will randomize subjects to lifestyle change or lifestyle change plus GLP-1 receptor agonist. Lifestyle change will be developed around a meal replacement strategy. The intervention will be weight loss using Slim-Fast®. Participants will be provided Slim-Fast® meal replacement shakes to utilize for two meals daily plus one to two 100 calorie snacks, similar to the Look AHEAD protocol. The subjects will receive specific menus and training on food composition to prepare one healthy 500 calorie meal daily, for a net hypocaloric diet.
  Interventions: Behavioral: Weight loss
- Weight loss plus liraglutide (Active Comparator): Patients will be randomized to lifestyle change and the GLP-1 agonist, liraglutide. Subjects in this group will be administered 0.6mg liraglutide, sq injection daily for 1 week, increased to 1.2 mg for 1 week, and then 3.0 mg for the next 10 weeks of the acute phase. This gradual escalation of the dose is designed to minimize gastrointestinal side effects. Empty syringes will be monitored for compliance.
  Interventions: Drug: Liraglutide; Behavioral: Weight loss

INTERVENTIONS:
Drug: Liraglutide — Active comparator. See arm descriptions.
  Other Names: Saxenda
  Arms: Weight loss plus liraglutide
Behavioral: Weight loss — Active comparator. See arm descriptions.

SUMMARY:
This study will examine the benefits of weight loss alone or in combination with a GLP1 receptor agonist, liraglutide, on beta cell function in young adult Mexican American (MA) women with prediabetes. The Investigators have chosen to focus on MA women because MA women are at very high risk for progression to diabetes and have not traditionally been involved in weight management studies since they are thought to be difficult to recruit and retain in such programs. However, investigators have had particular success in working with young MA women using specifically developed ethnic and gender conscious programs. Because weight loss does not prevent all progression to diabetes, some participants will receive the diabetes medication, liraglutide, which has been shown to stabilize beta cell function. The study will also interrogate for polymorphisms of known T2DM genes to correlate with beta cell response to weight loss and liraglutide treatment. Additionally, this investigation targets serious health disparities in metabolic disease in a highly vulnerable, rapidly growing population, testing novel gender and culturally focused intervention strategies and identifying genetic biomarkers of response to a pharmacologic intervention that targets the pancreatic ßcell.

These results will help to a) understand mechanisms of disease, b) personalize treatment through identification of a high risk group that may be amenable to specific therapy, and c) ultimately, sets the stage for an intervention trial to prevent diabetes, a major chronic and costly disease, in Mexican Americans.

DETAILED DESCRIPTION:
Investigators will test the hypothesis that liraglutide, because of its actions on the β-cell, will amplify the effects of lifestyle management to improve β-cell function. Investigators will recruit MA ages 18-40, since above this age the incidence of T2DM in obese MA women in our experience approaches 50%. The primary endpoint will be β-cell function (AIRg) in response to lifestyle change with and without GLP-1 agonist at 3 months. Secondary endpoints will be reversal of metabolic syndrome and changes in plasma biomarkers. By the end of 3 months, the prediabetic subject will be in the best possible metabolic control, and investigators would predict that the liraglutide group would reveal better β-cell function. Thus, data from this time point will be used for pharmacogenetic studies. The program will be continued for 3 more months for transition to regular healthy meals with the goal of weight maintenance. During this second 3 months, subjects will be off liraglutide to determine the sustainability of the improved β-cell function. In the absence of weight re-gain, investigators predict that the intensive weight loss alone group would maintain improved β-cell function, but the intensive weight loss+liraglutide group would display even better function. These results will provide useful information about improving β-cell function in the management of young women with pre-diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Mexican-american
* Female
* BMI 30-42
* willingness to complete protocol
* pre-diabetic
* English or Spanish literate

Exclusion Criteria:

* pregnant
* 30 min or more of moderate to vigorous activity more than 3 times per week
* cardiovascular disease
* physical limitations that might be aggravated by moderate physical activity
* planning to move in next 12-24 months
* diabetic

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2016-05; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Beta Cell Function | 3 months
  disposition index: x10^-5min-1

SECONDARY OUTCOMES:
Waist Circumference | 3 months
  inches
Fasting Glucose | 3 months
  mg/dL
Triglycerides | 3 months
  mg/dL
HDL cholesterol | 3 months
  mg/dL
Blood Pressure | 3 months
  mmHg
Heart Sensitive C-reactive protein | 3 months
  hsCRP, mg/L
Presence of genetic polymorphisms | 3 months
  yes or no

CONTACTS AND LOCATIONS:
Overall Officials: David Bradley, MD, Principal Investigator — Ohio State University
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - L.A. Biomedical Research Institute, Torrance, California
  - Magnolia Multiservice Center, Houston, Texas
  - Denver Harbor Multi-service Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Publication, presentation

REFERENCES:
- [Background] Hsueh WA, Orloski L, Wyne K. Prediabetes: the importance of early identification and intervention. Postgrad Med. 2010 Jul;122(4):129-43. doi: 10.3810/pgm.2010.07.2180. PMID 20675976
- [Background] Bergman RN, Ader M, Huecking K, Van Citters G. Accurate assessment of beta-cell function: the hyperbolic correction. Diabetes. 2002 Feb;51 Suppl 1:S212-20. doi: 10.2337/diabetes.51.2007.s212. PMID 11815482
- [Background] Matveyenko AV, Butler PC. Relationship between beta-cell mass and diabetes onset. Diabetes Obes Metab. 2008 Nov;10 Suppl 4(0 4):23-31. doi: 10.1111/j.1463-1326.2008.00939.x. PMID 18834430
- [Background] Villareal DT, Banks MR, Patterson BW, Polonsky KS, Klein S. Weight loss therapy improves pancreatic endocrine function in obese older adults. Obesity (Silver Spring). 2008 Jun;16(6):1349-54. doi: 10.1038/oby.2008.226. Epub 2008 Apr 3. PMID 18388888
- [Background] Degn KB, Juhl CB, Sturis J, Jakobsen G, Brock B, Chandramouli V, Rungby J, Landau BR, Schmitz O. One week's treatment with the long-acting glucagon-like peptide 1 derivative liraglutide (NN2211) markedly improves 24-h glycemia and alpha- and beta-cell function and reduces endogenous glucose release in patients with type 2 diabetes. Diabetes. 2004 May;53(5):1187-94. doi: 10.2337/diabetes.53.5.1187. PMID 15111485
- [Background] Mari A, Degn K, Brock B, Rungby J, Ferrannini E, Schmitz O. Effects of the long-acting human glucagon-like peptide-1 analog liraglutide on beta-cell function in normal living conditions. Diabetes Care. 2007 Aug;30(8):2032-3. doi: 10.2337/dc07-0310. Epub 2007 Apr 27. No abstract available. PMID 17468345
- [Background] Look AHEAD Research Group; Wing RR. Long-term effects of a lifestyle intervention on weight and cardiovascular risk factors in individuals with type 2 diabetes mellitus: four-year results of the Look AHEAD trial. Arch Intern Med. 2010 Sep 27;170(17):1566-75. doi: 10.1001/archinternmed.2010.334. PMID 20876408
- [Background] Goodarzi MO, Taylor KD, Scheuner MT, Antoine HJ, Guo X, Shah PK, Rotter JI. Haplotypes in the lipoprotein lipase gene influence high-density lipoprotein cholesterol response to statin therapy and progression of atherosclerosis in coronary artery bypass grafts. Pharmacogenomics J. 2007 Feb;7(1):66-73. doi: 10.1038/sj.tpj.6500402. Epub 2006 Jun 6. PMID 16755277
- [Background] Krauss RM, Mangravite LM, Smith JD, Medina MW, Wang D, Guo X, Rieder MJ, Simon JA, Hulley SB, Waters D, Saad M, Williams PT, Taylor KD, Yang H, Nickerson DA, Rotter JI. Variation in the 3-hydroxyl-3-methylglutaryl coenzyme a reductase gene is associated with racial differences in low-density lipoprotein cholesterol response to simvastatin treatment. Circulation. 2008 Mar 25;117(12):1537-44. doi: 10.1161/CIRCULATIONAHA.107.708388. Epub 2008 Mar 10. PMID 18332269
- [Background] Mangravite LM, Medina MW, Cui J, Pressman S, Smith JD, Rieder MJ, Guo X, Nickerson DA, Rotter JI, Krauss RM. Combined influence of LDLR and HMGCR sequence variation on lipid-lowering response to simvastatin. Arterioscler Thromb Vasc Biol. 2010 Jul;30(7):1485-92. doi: 10.1161/ATVBAHA.110.203273. Epub 2010 Apr 22. PMID 20413733